CLINICAL TRIAL: NCT07238140
Title: Comparative Study Between Automatic Tube Compensation and Pressure Support Ventilation as a Mode of Weaning From Mechanical Ventilation in Patients With Respiratory Failure
Brief Title: ATC vs PSV for Weaning in Patients With Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Kamal Habib, Lecturer of Anesthesia and Intensive Care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMASU MS 69/2019
Record Dates: First submitted 2025-10-01; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: weaning; ATC; PSV
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated into two parallel groups: ATC group and PSV group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATC group (Experimental): ATC mode was applied at 100% compensation during the spontaneous breathing trial using a Puritan-Bennett 840 ventilator. Patients breathed through the ventilator circuit with flow triggering (1 L/min), PEEP of 5 cmH₂O, and FiO₂ < 0.5. This intervention aimed to assist patients during weaning from mechanical ventilation.
  Interventions: Device: Automatic tube compensation
- PSV Group (Active Comparator): Patients were weaned using Pressure Support Ventilation (PSV). They breathed through the ventilator circuit with flow triggering (1 L/min), PEEP of 5 cmH₂O, FiO₂ < 0.5, and pressure support adjusted to achieve a tidal volume of 6-8 mL/kg predicted body weight.
  Interventions: Device: Pressure Support Ventilation

INTERVENTIONS:
Device: Automatic tube compensation — Automatic Tube Compensation (ATC) mode was applied at 100% using a Puritan-Bennett 840 ventilator during spontaneous breathing trials. This mode compensates for the additional resistance imposed by the endotracheal tube, thereby reducing patients' work of breathing and facilitating weaning from mechanical ventilation. Flow triggering was set at 1 L/min, with PEEP of 5 cmH₂O and FiO₂ < 0.5.
  Other Names: ATC
  Arms: ATC group
Device: Pressure Support Ventilation — Pressure Support Ventilation (PSV) was applied during spontaneous breathing trials using a Puritan-Bennett 840 ventilator. Patients breathed through the ventilator circuit with flow triggering set at 1 L/min, positive end-expiratory pressure (PEEP) of 5 cmH₂O, and fraction of inspired oxygen (FiO₂) < 0.5. Pressure support levels were adjusted to achieve a tidal volume of 6-8 mL/kg of predicted body weight
  Other Names: PSV
  Arms: PSV Group

SUMMARY:
Comparative study between automatic tube compensation and pressure support ventilation as a mode of weaning from mechanical ventilation in patients with respiratory failure

DETAILED DESCRIPTION:
Mechanical ventilation is a cornerstone in the management of patients with acute respiratory failure, but prolonged dependence on the ventilator is associated with increased morbidity, mortality, and healthcare costs. Weaning, the process of transitioning a patient from mechanical ventilation to spontaneous breathing, is a critical phase that requires careful timing and appropriate methodology. The spontaneous breathing trial (SBT) is a widely used tool to assess weaning readiness, and several ventilatory modes have been developed to optimize this step. Among these, Automatic Tube Compensation (ATC) and Pressure Support Ventilation (PSV) are two commonly applied modes, each with distinct physiological principles.

ATC is designed to compensate precisely for the resistance imposed by the endotracheal tube, aiming to reproduce the normal work of breathing as if the patient were breathing without the artificial airway. In contrast, PSV provides a fixed level of pressure support throughout inspiration, which assists respiratory muscles and reduces the work of breathing but may not adapt dynamically to changes in flow or resistance. Although both modes are frequently used in intensive care units, evidence comparing their effectiveness in facilitating weaning and extubation success has been variable, with some studies suggesting physiological advantages of ATC but limited data on clinical outcomes.

his prospective randomized clinical trial was conducted to address this gap by directly comparing ATC and PSV as SBT modes in adult patients with acute respiratory failure receiving invasive mechanical ventilation. Patients were screened for weaning readiness using standardized clinical and physiological criteria and were subsequently randomized to undergo SBT with either ATC or PSV. Interventions were delivered following established ICU protocols to ensure safety and uniformity across groups.

Throughout the study, key respiratory and gas exchange parameters were monitored before and after the SBT to assess physiological responses to the two modes. Extubation decisions were based on predefined criteria to minimize variability in clinical judgment. Patients were followed for early post-extubation outcomes to evaluate the clinical impact of each mode on weaning success. The primary endpoint focused on improvement in oxygenation, while secondary endpoints included respiratory mechanics and post-extubation outcomes. The study adhered to ethical regulations, with written informed consent obtained prior to enrollment. By providing a structured comparison of these two modes, the study contributes to the evidence guiding optimal weaning strategies in adult critically ill patients, potentially improving clinical outcomes and optimizing ICU resource utilization.

Statistical analysis was performed using SPSS software (version 16.0; IBM Corp., Armonk, NY, USA). The required sample size was calculated a priori to provide 80% power to detect a clinically meaningful difference in the primary outcome at a two-sided significance level of 0.05. Continuous variables were expressed as mean ± standard deviation and compared between groups using appropriate parametric tests. Categorical variables were presented as frequencies and percentages, and analyzed using the Chi-square test or Fisher's exact test as indicated. A P value < 0.05 was considered statistically significant. Diagnostic accuracy was assessed using receiver operating characteristic (ROC) curve analysis, with calculation of sensitivity, specificity, positive predictive value, and negative predictive value.

The results of this completed study provide valuable clinical evidence regarding the optimal mode of spontaneous breathing trials in adult patients with acute respiratory failure. By comparing ATC and PSV, the study highlights differences in physiological responses and clinical outcomes between the two modes. These findings can help refine weaning protocols, support clinical decision-making, and contribute to improving extubation success rates and patient outcomes in intensive care settings. Moreover, the results may serve as a reference for future research and guideline development, particularly in resource-limited environments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Admitted with acute respiratory failure (ARF).
* On mechanical ventilation with Puritan-Bennett 840 ventilator for ≥24 hours.
* Considered for weaning after improvement or resolution of underlying cause.
* Fully conscious.
* Minimal or no requirement for vasoactive drugs or sedation.
* Adequate gas exchange (PaO₂/FiO₂ >200 at PEEP 5 cmH₂O and FiO₂ <0.5) Rapid shallow breathing index (RSBI) <105 breaths/min/L.

Exclusion Criteria:

* Age <18 years.
* Pre-existing chronic obstructive pulmonary disease (COPD).
* Neuromuscular disorders.
* Hemodynamic instability requiring high-dose vasoactive support.
* Persistent altered level of consciousness.
* Ongoing sedation.
* Severe metabolic or electrolyte disturbances.
* Morbid obesity (BMI ≥40 kg/m²).
* Tracheostomy.
* Pregnancy.
* Refusal to participate by patient or legal guardian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-26 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Change in PaO₂/FiO₂ ratio (oxygenation index) during spontaneous breathing trial | Immediately before and at the end of the spontaneous breathing trial (SBT), assessed up to 2 hours
  The primary outcome was the change in the PaO₂/FiO₂ ratio measured immediately before and at the end of the spontaneous breathing trial (SBT). This parameter reflects the efficiency of oxygen exchange and is a validated predictor of weaning success. Higher improvements in the PaO₂/FiO₂ ratio indicate better respiratory function and a higher likelihood of successful extubation.

SECONDARY OUTCOMES:
Change in Respiratory Rate to Tidal Volume Ratio (RR/VT) | Immediately before and at the end of the spontaneous breathing trial (SBT), assessed up to 2 hours
  Assessment of the rapid shallow breathing index (RR/VT) as a predictor of weaning success. Measurements will be taken at baseline and at the end of the spontaneous breathing trial to assess changes during weaning.
Change in Oxygen Saturation (SpO₂) | Immediately before and at the end of the spontaneous breathing trial (SBT), assessed up to 2 hours
  Evaluation of oxygen saturation changes during the spontaneous breathing trial to assess the patient's oxygenation status.
Change in Dynamic Compliance | Immediately before and at the end of the spontaneous breathing trial (SBT), assessed up to 2 hours
  Measurement of dynamic respiratory system compliance to assess lung mechanics before and after the spontaneous breathing trial.
Change in Airway Resistance | Immediately before and at the end of the spontaneous breathing trial (SBT), assessed up to 2 hours
  Assessment of changes in airway resistance during weaning to evaluate respiratory mechanics at baseline and after the SBT
Change in Intrinsic PEEP | Immediately before and at the end of the spontaneous breathing trial (SBT), assessed up to 2 hours
  Measurement of intrinsic PEEP values before and after the spontaneous breathing trial to assess changes in auto-PEEP during weaning.
Change in Arterial Oxygen Tension (PaO₂) | Immediately before and at the end of the spontaneous breathing trial (SBT), assessed up to 2 hours
  Assessment of PaO₂ changes during weaning to evaluate oxygenation efficiency before and after the spontaneous breathing trial.
Change in Arterial Carbon Dioxide Tension (PaCO₂) | Immediately before and at the end of the spontaneous breathing trial (SBT), assessed up to 2 hours
  Assessment of PaCO₂ changes during weaning to evaluate ventilation efficiency before and after the spontaneous breathing trial.
Extubation Success Rate | Up to 48 hours post-extubation
  Proportion of patients who maintain spontaneous breathing without signs of respiratory distress or hemodynamic instability for 48 hours after extubation. This outcome assesses the overall success of weaning.

CONTACTS AND LOCATIONS:
Locations (1):
- intensive care unit Department, Ain Shams University Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study, including clinical parameters, ventilatory settings, oxygenation indices, and demographic information, will be shared with qualified researchers upon request after publication of the study results. Requests will be reviewed by the Principal Investigator, and approved data will be shared via a secure repository. No personal identifiers will be included to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: * Start Date: Upon publication of the study results.
  * End Date: 5 years after publication.
Access Criteria: Qualified researchers may request access to de-identified individual participant data (IPD) from this study, including clinical parameters, ventilatory settings, oxygenation indices, and demographic information. Supporting information such as Study Protocol, Statistical Analysis Plan (SAP), and Clinical Study Report (CSR) will also be provided. Requests will be submitted to the Principal Investigator for review. Approved requests will receive the data through a secure repository to ensure confidentiality. Data will not include any personal identifiers, and access is limited to research purposes only.